CLINICAL TRIAL: NCT04998721
Title: A Dyadic Approach to Perinatal Depression in Primary Care: Maternal Infant and Dyadic Care (MInD)
Brief Title: A Dyadic Approach to Perinatal Depression in Primary Care: Maternal Infant and Dyadic Care
Acronym: MInD
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: University of Washington (Other)
Collaborators: National Institute of Mental Health (NIMH) (NIH)
Responsible Party: Principal Investigator, Amritha Subray Bhat, Assistant Professor, School of Medicine: Psychiatry, University of Washington
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: STUDY00011405; 1R34MH124798-01 (NIH)
Record Dates: First submitted 2021-07-22; First posted 2021-08-10 (Actual); Last update posted 2023-12-22 (Actual); Status verified 2023-11

CONDITIONS: Depression, Postpartum; Efficacy, Self; Anxiety
MeSH Terms: conditions — Depression, Postpartum; Anxiety Disorders

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Maternal Infant Dyadic Care (Experimental): Perinatal collaborative care and Promoting First Relationships-Brief
  Interventions: Behavioral: Promoting First Relationships-Brief; Behavioral: Perinatal Collaborative Care
- Control (Active Comparator): Perinatal collaborative care only
  Interventions: Behavioral: Perinatal Collaborative Care

INTERVENTIONS:
Behavioral: Promoting First Relationships-Brief — A brief version of the evidence based Promoting First Relationships (PFR) parenting intervention in which a parent is supported in appropriate interpretation of infant cues and in developing skills to effectively parent an infant. Sessions consist of reflective content (observing and reflecting back to the mother on patterns of dyadic interaction) and informational handouts. Reflective content will be delivered in person, and text messaging protocol will deliver informational content at developmentally appropriate times. PFR-B sessions are delivered in primary care settings beginning in the third trimester and continuing postpartum.
  Arms: Maternal Infant Dyadic Care
Behavioral: Perinatal Collaborative Care — Collaborative Care (CC) is an integrated care model that is effective in the treatment of perinatal depression. CC provides team driven, population focused, measurement guided and evidence based care to improve access and outcomes, control costs, and increase patient satisfaction.

SUMMARY:
The purpose of this study is to assess the effectiveness of a parenting intervention+usual care compared to usual care on postpartum depression and other mental health and parenting outcomes, as well as the feasibility and acceptability of the parenting intervention.

DETAILED DESCRIPTION:
Eligible and consenting participants will be randomized in a single blind manner (research visitor will be blinded to condition) at a 1:1 ratio to either MInD (parenting intervention and usual perinatal collaborative care) or usual collaborative care in their second trimester of pregnancy. Research assessments will be administered during pregnancy and post-partum.

ELIGIBILITY:
Inclusion Criteria:

* English speaking pregnant women between gestational age (GA) 13 - 24 weeks
* ≥ 18 years,
* EPDS score ≥10,
* Ability to send and receive text messages (TM)

Exclusion Criteria:

* Severe substance use disorder in the past 6 months (score of 4 or above on the Alcohol Use Disorders Test AUDIT-C or a score of 6 or more on the Drug Abuse Screening Test (DAST).
* Active suicidal ideation as measured by follow up to a positive answer to question 10 on the EPDS.
* Bipolar disorder (Composite International Diagnostic Interview score ≥7) or psychotic disorder (assessed by chart review);
* Multiple gestation (assessed by self-report and medical record);
* Ongoing active treatment with psychotropic medications by mental health specialist (but not a PCP or Obstetrician).

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2022-11-01 (Actual); Primary Completion 2025-03-01 (Estimated); Study Completion 2025-06-01 (Estimated)

PRIMARY OUTCOMES:
Change from Baseline in Perinatal Depression Symptomology on the Edinburgh Postnatal Depression Scale (EPDS) | Baseline, 30-34 Weeks Gestational Age, 6 Weeks Postpartum, 3 Months Postpartum, 6 Months Postpartum
  The EPDS is a ten-item self-report depression measure with higher scores indicating increased symptoms severity, total score ranging from 0 to 30 and is validated for use in the perinatal period.

SECONDARY OUTCOMES:
Change from Baseline in Parental Self-Efficacy on the Self-Efficacy in a Nurturing Role (SENR) | Baseline, 30-34 Weeks Gestational Age, 6 Weeks Postpartum, 3 Months Postpartum, 6 Months Postpartum
  The SENR contains 16 items rated on 7-point scales regarding mothers' perceptions of their competence on basic skills required in caring for an infant (e.g., "I feel confident in my role as a parent," "I can soothe my baby easily when he or she is crying or fussing") In the prenatal assessment questions address how women expect to do once their infant is born (e.g., "I look forward to becoming a parent with confidence in my role as a parent," "I expect to be able to soothe my baby easily when he or she is crying or fussing"). Scores on the SENR are obtained by summing individual items to yield a total efficacy score, with higher scores reflecting greater feelings of efficacy.
Change from Postpartum Baseline in Dyadic Interaction | 6 Weeks Postpartum, 3 Months Postpartum, 6 Months Postpartum
  Dyadic interaction will be coded using the NCAST applied to mother and child interactive behavior during a 3-minute videotaped session.
Change from Baseline in Disability on the World Health Organization Disability Assessment Schedule 2.0 (WHODAS) | Baseline, 30-34 Weeks Gestational Age, 6 Weeks Postpartum, 3 Months Postpartum, 6 Months Postpartum
  WHODAS 2.0 is a 12 item assessment of overall functioning. The scores assigned to each of the items - "none" (0), "mild" (1) "moderate" (2), "severe" (3) and "extreme" (4) - are summed, total score ranging from 0 to 48.
Change from Postpartum Baseline in Maternal Functioning on the Barkin Index of Maternal Functioning (BIMF) | 6 Weeks Postpartum, 3 Months Postpartum, 6 Months Postpartum
  The BIMF is a 20-item self-report measure for use in the first year postpartum and can assess overall functioning in the context of new motherhood. It measures the functional domains of social support, management, mother-child interaction, infant care, self-care, adjustment, and psychological well-being (of the mother). It is measured only postpartum. A total score is generated from summing the 20 items and ranges from 0 to 120.
Relative utilization of MInD vs usual CC | Baseline through up to 6 Months Postpartum (up to maximum of 9 months)
  The investigators operationalize adequate treatment utilization as participating in a sufficient number of health care encounters to achieve a therapeutic effect: attendance at ≥6 care manager sessions (≥3 prenatal and ≥3 postpartum).
Perceived match of treatment to patient need using Working Alliance Inventory (WAI-SR) | 30-34 Weeks Gestational Age, 6 Weeks Postpartum, 3 Months Postpartum, 6 Months Postpartum
  The investigators will administer the Working Alliance Inventory (WAI-SR) to all enrolled women to assess strength of alliance with the therapist and compare mean change over time between MInD and usual CC groups.

CONTACTS AND LOCATIONS:
Overall Officials: Amritha S Bhat, MD, MPH, Principal Investigator — University of Washington
Locations (1):
- Amritha Bhat, Seattle, Washington, United States